CLINICAL TRIAL: NCT06296758
Title: Femoral Nerve Blockade (FNB) vs Suprainguinal Fascia Iliaca Block (SiFi) for Hip Fracture Surgery
Brief Title: SiFi vs FNB Local Anesthesia for Hip Fracture Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SiFi_HIP FRACTURE
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hip Fractures; Surgery; Anesthesia, Local
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: A concealed-allocation parallel-group blinded randomized controlled clinical
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be conducted through blocked randomization with blocks of 4 according to a schedule not known to the investigators using a computerized algorithm. The attending surgeon, anesthetist, and nursing team will be blinded to the randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIFI local anesthesia (Experimental): Subjects randomized to the SiFi arm will have an ultrasound-guided suprainguinal fascia iliaca single shot block performed preoperatively in the anesthesia block room with 40ml of 0.2% ropivacaine local anesthetic. This will be reduced to 30 ml in patients under 60 kg.
  Interventions: Procedure: Regional anesthesia
- FNB local anesthesia (Active Comparator): Subjects randomized to the FNB arm will have an ultrasound-guided femoral nerve single shot block performed preoperatively in the anesthesia block room with 20ml of 0.5% ropivacaine local anesthetic. This will be reduced to 15ml in patients under 60 kg.
  Interventions: Procedure: Regional anesthesia

INTERVENTIONS:
Procedure: Regional anesthesia — ultrasound-guided suprainguinal fascia iliaca block with 40ml of ropivacaine local or ultrasound-guided femoral nerve block with 20ml of ropivacaine local anesthetic

SUMMARY:
The goal of this clinical trial is to compare two commonly used local/regional anesthesia techniques in adults patients undergoing hip fracture surgery. The main question[s] it aims to answer are: • the impact of both interventions on patient level of pain. • impact on postoperative analgesics administered Participants will be randomly assigned to one of two local/regional anesthesia techniques, either femoral nerve block (FNB) or suprainguinal fascia iliaca block (SiFi). Both techniques are the usual practice at the hospital, and we are NOT aiming to experiment on new anesthesia technique in this study.

DETAILED DESCRIPTION:
Hip fracture in the elderly is an increasingly common problem worldwide. Nearly all patients with a hip fracture undergo surgery. Patients with hip fractures often have significant pain, particularly with movement, and surgical fixation is associated with significant pain.

The treatment of pain with the use of a multimodal analgesic regimen is a major priority for elderly patients with hip fractures. These patients are often frail and have multiple medical comorbidities. Hence the use of non-steroidal anti-inflammatories drugs and systemic opioids may be contraindicated or complicated by adverse effects. Regional anesthesia techniques including femoral nerve blocks (FNB) and fascia iliaca compartment blocks (FICB) are frequently utilized as part of multimodal analgesia due to their relative lack of side-effects. Femoral nerve blockade and suprainguinal fascia iliaca (SiFi) blockade have been described for this indication. Several studies have investigated the analgesic efficacy of the SiFi block after total hip arthroplasty. However, randomized controlled trials on the analgesic efficacy of the SiFi block for pain after hip fracture surgery are not plentiful and subject to methodological concerns.

Objectives:

The primary objective is to test the hypothesis that in patients undergoing hip fracture surgery, suprainguinal fascia iliaca block is associated with improved pain scores and a reduction in opioid utilization when compared with femoral nerve block. Secondary objectives will be to compare time to mobilization, time to readiness for discharge and complications associated with both nerve block techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Having hip fracture surgery at the University of Alberta Hospital
* Suitable for multimodal analgesia including a peripheral nerve block

Exclusion Criteria:

* Contraindication to a nerve block technique
* Refuses consent for a nerve block technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours
  Postoperative numerical pain rating scale (NRS) pain scores
Postoperative analgesics administered | 48 hours
  Postoperative opioid utilization

SECONDARY OUTCOMES:
Mobilization | 48 hours
  Time to first mobilization
Time to readiness for discharge | 48 hours
  Time to 'ready for discharge'
Complications | 48 hours
  Complications associated with both block techniques

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make the individual participants data available to other researchers was made